CLINICAL TRIAL: NCT01140516
Title: Antibiotic prophyLaxis Versus Placebo in Infants Diagnosed With Hydronephrosis Antenatally
Brief Title: Effectiveness of Antibiotics Versus Placebo to Treat Antenatal Hydronephrosis
Acronym: ALPHA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: McMaster University (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other); Hamilton Health Sciences Corporation (Other); McMaster Surgical Associates (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALPHA
Record Dates: First submitted 2010-06-08; First posted 2010-06-09 (Estimated); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Hydronephrosis; Urinary Tract Infection
Keywords: Antenatal
MeSH Terms: conditions — Hydronephrosis; Urinary Tract Infections | interventions — Trimethoprim

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Trimethoprim (Active Comparator): Prophylactic Antibiotics
  Interventions: Drug: Trimethoprim
- Simple syrup (Placebo Comparator): 2mg/kg,orally until febrile UTI occurs or until completion of the study if the patients do not develop any UTI.
  Interventions: Other: Simple Syrup

INTERVENTIONS:
Drug: Trimethoprim — 2mg/kg,orally until febrile UTI occurs or until completion of the study if the patients do not develop any UTI.
  Arms: Trimethoprim
Other: Simple Syrup — 2mg/kg,orally until febrile UTI occurs or until completion of the study if the patients do not develop any UTI.
  Arms: Simple syrup

SUMMARY:
This study focuses on the relationship between prophylaxis antibiotics and frequency of urinary tract infection in children diagnosed with antenatal hydronephrosis. Hydronephrosis is the most common fetal abnormality occurring in 1-5% of all pregnancies. Currently, with the widespread accessibility of antenatal ultrasound across cities in Ontario, the detection of hydronephrosis has become even more common. As a result, thousands of infants with hydronephrosis have been seen and managed by pediatricians, pediatric nephrologists, pediatric urologists, and family physicians. The investigators need to determine if antibiotic prophylaxis is effective in reducing the number of urinary tract infections in this population.

DETAILED DESCRIPTION:
This study focuses on the relationship between prophylaxis antibiotics and frequency of urinary tract infection in children diagnosed with antenatal hydronephrosis. Hydronephrosis is the most common fetal abnormality occurring in 1-5% of all pregnancies. Currently, with the widespread accessibility of antenatal ultrasound across cities in Ontario, the detection of hydronephrosis has become even more common. As a result, thousands of infants with hydronephrosis have been seen and managed by pediatricians, pediatric nephrologists, pediatric urologists, and family physicians. The investigators need to determine if antibiotic prophylaxis is effective in reducing the number of urinary tract infections in this population.To determine whether CAP reduces the rate of UTI in infants with prenatal HN within the first 18 months of life.

This is superiority, parallel, blinded, randomized, placebo-controlled trial in infants with prenatal HN testing the effect of CAP on febrile UTI rates over the first 18 months of life

For clinical and safety purposes, data will be collected on symptoms and signs of febrile laboratory confirmed UTI (urinalysis, urine culture), compliance to treatment, adverse effects, and resistance to prophylactic antibiotics in case of positive urine cultures. As part of standard medical care, the patient and family are scheduled for renal-bladder ultrasounds and outpatient pediatric urology clinic visits at the local recruitment sites (i.e. McMaster Children's Hospital, The Hospital for Sick Children or, Children's Hospital of Eastern Ontario) during months as mentioned above at baseline, 3, 6, 9 and 12 months . During these clinic appointments, the research coordinator will follow up with patient and family regarding their progress in the study. The Research Coordinator will ask about any side effects from trial medication (nausea, vomiting, gastroenteritis, anaphylactic reactions) and ensure their questions or concerns are addressed. Data from patient's ultrasound assessment and renal scans will also be collected.

In addition to clinic follow ups, patients and their families will be contacted monthly (excluding the months patient is scheduled for clinical follow up) by the Research Coordinator to further monitor patient's study progress. Families will be instructed to call the Research Coordinator at the first sign of febrile UTI (fever, loss of appetite, abdominal pain) and advised to seek medical assistance (bring their child to the Emergency Department at the local study institution). The baby will then have a dipstick taken to test for positive nitrites and leukocytes. If positive, patients are to have a urine sample via catheter specimen taken and if positive, be taken off study medication and be treated for febrile UTI according to standard medical practice. In this case the family and healthcare providers will not be unblinded to the participant's treatment allocation as this information is not required in order to treat the infant. In the event that parents are unable to bring their child to the local study institution, it is advised they obtain a dipstick and a catheter specimen from their local walk-in-clinic, Urgent Care Centre or family physician's office. If a catheter specimen is not available at these locations, a sterile bag may be used to determine outcome of urine sample. To ensure there is consistency between outside facilities, parents are given detailed instructions to obtain a dipstick and provide a photocopy of the results to the Research Coordinator for our records and potential adjudication.

Letters will be faxed to the doctor that treated the child for the suspected UTI in order to obtain the associated reports.

ELIGIBILITY:
Inclusion Criteria:

1. Infants with AHN (one to seven months of age) confirmed postnatally with renal-bladder ultrasound and/or a dilated ureter ≥ 7mm
2. SFU grade III and IV AHN (high grade hydronephrosis)
3. Patients without grades II to V VUR determined by voiding cystogram (includes UPJO-like and primary megaureter (hydroureteronephrosis) only);
4. Parent or legal guardian able to give free and informed consent

Exclusion Criteria:

1. Infants with grades II to V VUR
2. Infants with posterior urethral valves or Prune-Belly syndrome
3. Duplication anomalies (ureteroceles, ectopic ureters)
4. Other conditions that may require chronic use of antibiotics
5. Previous renal failure
6. Allergy to trimethoprim
7. Co-enrollment in another intervention trial

Ages: 1 Month to 7 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Estimated)
Dates: Start 2010-07; Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
To determine whether antibiotics (ATB) prophylaxis prevents urinary tract infection (UTI) in infants with antenatal hydronephrosis (AHN). | The outcome measures will be assessed at 12 months
  Determine the rate and frequence of UTI infection

CONTACTS AND LOCATIONS:
Overall Officials: Luis H Braga, MD, MSc, PhD, Principal Investigator — McMaster Medical Centre, McMaster University
Locations (2):
- Canada (2):
  - McMaster Children's Hospital, Hamitlon, Ontario
  - Sick Kids Hospital for Sick Children, Toronto, Ontario